CLINICAL TRIAL: NCT05884489
Title: Gamified Smartphone Application to Improve the Adherence to the Mediterranean Diet in Cardiac Patients: a Usability and Feasibility Study
Brief Title: Usability and Feasibility of the NutriQuest Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022/058
Record Dates: First submitted 2023-05-09; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Gamification; Nutrition; Behavior Change
Keywords: Gamification; Smartphone; Mediterranean diet; Nutrition; Cardiovascular diseases; Intervention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Behavioral: A gamified smartphone app-based eating behaviour intervention

INTERVENTIONS:
Behavioral: A gamified smartphone app-based eating behaviour intervention — All patients gained access to the healthy nutrition application and were encouraged to make full use of its feature, and they were also required to maintain a logbook through the application at home to follow-up on their diet. The intervention last for six weeks.

SUMMARY:
The study is a pilot study (phase 2) that includes a usability study (phase 1).

The aim of the study is to investigate the feasibility and usability of the healthy nutrition application and the effects on adherence to Modified Mediterranean diet, self-efficacy and nutrition knowledge among patients with cardiovascular disease in a cardiac rehabilitation setting. Furthermore, it studies the overall user experience when using the healthy nutrition application.

DETAILED DESCRIPTION:
The study can be divided in two phases, each one addressing a specific research question:

1. Usability: Is the developed healthy nutrition application user-friendly and does it seem motivating for cardiac patients in a cardiac rehabilitation setting to use the application to eat more healthily?
2. Pilot study: Is the developed healthy nutrition application feasible and acceptable for cardiac patients? Does the healthy nutrition application have an effect on adherence to Modified Mediterranean diet, self-efficacy and nutrition knowledge in cardiac patients in a cardiac rehabilitation setting and what is the user experience?

ELIGIBILITY:
Inclusion Criteria:

* History of cardiovascular disease with or without intervention (PCI/CABG/conservative/pacemaker implantation/ablation)
* History of current or past cardiac rehabilitation in Jessa Hospital Hasselt
* Current treatment must require them to follow the Mediterranean diet plan
* Age ≥18 years
* Willing and physically able to follow a application-based healthy nutrition program and other study procedures in a six-week follow-up period
* Evidence of a personally signed and dated informed consent, indicating that the subject (or a legally-recognized representative) has been informed of all pertinent aspects of the study
* Possession of and/or able to use an Android based smartphone (version 6 or higher)
* Possession of internet connectivity
* Dutch speaking and understanding

Exclusion Criteria:

* Pregnant females
* Combined with diabetes or severe kidney disease
* Participation in other cardiac rehabilitation program trials, focusing on diet outcome
* Current or recent participation in other technology-supported programs, even when not directly targeting nutrition
* Any condition which in the opinion of the investigator would make it unsafe or unsuitable for the patient to participate in this study or a life expectancy of less than six weeks based on investigators judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Usability | Six week
  The usability questionnaire asks patients to evaluate various components of the application based on perceived usefulness, ease of use and ease of understanding, as well as visual attractiveness and contains various questions specific to each component. The questionnaire includes 109 questions, we use 5-point Likert scale. The higher score means better usability.
Motivation | Six week
  Motivation is measured by Intrinsic Motivation Inventory(IMI), it includes 18 items, we use 5-point Likert scale, the scores range from 18 to 90. Higher score means higher motivation.
Application visits | During the whole six week
  Usability is also measured by the objective index "application visits", the visits to each page/component of the application during the whole six week are recorded in the application.
Acceptance | Six week
  The acceptance is measured by Self-reported habit index(SRHI). It includes 12 items, we use 7-point Likert scale. Scores ranged from 12 to 84. The higher the score, the higher the acceptability.

SECONDARY OUTCOMES:
Change from baseline Adherence to Mediterranean diet at 6 weeks | Baseline and six week
  The adherence to Mediterranean diet is measured by Modified MedDietScore(MMDS), the MMDS we used in this study is an adaption of the MedDietScore in which parameters about salt and sugar intake are added to the score, and an intake of zero alcohol is considered positive (in contrast to the MedDietScore, which allows limited alcohol consumption), the higher score means better adherence to Mediterranean diet.
Change from Self-efficacy at 6 weeks | Baseline and Six week
  Self-efficacy is measured by "Nutrition self-efficacy scale", it includes five items, response format is (1) very uncertain, (2) rather uncertain, (3) rather certain, and (4) very certain. The higher the score indicates better self-efficacy.
Change from Knowledge at 6 weeks | Baseline and six week
  Knowledge is measured by "Nutrition knowledge score",the questionnaire contains 14 questions used to examine patients' knowledge about a healthy diet. Each question (e.g., what nutrients do not contain energy?) has four possible responses (e.g., proteins, alcohol, carbohydrates and minerals) and patients are expected to select the correct one. A question is worth one point, the higher the score indicates better nutrition knowledge.
Digital health literacy | Baseline
  The questionnaire includes five subscales (i.e. digital usage, digital skills, digital literacy, digital health literacy, and digital learnability) measured by 20 items that are answered on a 5-point Likert scale ranging from 1 to 5. Digital health literacy scores are calculated based on the sum of the four first subscales. The minimum score of the DHRQ is 15, and the maximum is 75. The score of digital learnability ranges from 5 to 25 and was categorized into 4 groups A (21-25), B (16-20), C (11-15), and D (5-10). Higher scores indicate greater willingness to learn about digital health tools. The result can be communicated as the total score + the letter from the digital learnability.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department, Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No